CLINICAL TRIAL: NCT02221752
Title: Impact of Iron/Folic Acid Versus Folic Acid Supplements During Pregnancy on Maternal and Children's Health: A Randomized Controlled Trial in China
Brief Title: Impact of Iron/Folic Acid vs Folic Acid Supplements During Pregnancy on Maternal and Child Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhao gengli (Other)
Collaborators: Vifor Pharma (Industry)
Responsible Party: Sponsor-Investigator, Zhao gengli, Associate Professor, Peking University First Hospital
Organization: Peking University First Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Vifor/PFH supplement trial
Record Dates: First submitted 2014-08-18; First posted 2014-08-20 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Iron Deficiency; Iron Deficiency Anemia
Keywords: iron deficiency; iron deficiency anemia; infant; pregnancy
MeSH Terms: conditions — Iron Deficiencies; Anemia, Iron-Deficiency | interventions — ferrous sulfate; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Folic acid (Experimental): Mothers randomized to receive 2 capsules per day: one with placebo and one with 0.40 mg folic acid from enrollment to delivery.
  Interventions: Dietary Supplement: Folic acid
- Ferrous Sulfate + folic acid (Experimental): Mothers randomized to receive 2 capsules per day: one with iron (300 mg ferrous sulfate [60 mg elemental iron]) and the other with 0.40 mg folic acid from enrollment to delivery.
  Interventions: Dietary Supplement: Ferrous Sulfate + folic acid

INTERVENTIONS:
Dietary Supplement: Ferrous Sulfate + folic acid — Mothers randomized to receive 2 capsules per day: one with iron (300 mg ferrous sulfate [60 mg elemental iron]) and the other with 0.40 mg folic acid from enrollment to delivery.
  Arms: Ferrous Sulfate + folic acid
Dietary Supplement: Folic acid — Mothers randomized to receive 2 capsules per day: one with placebo and one with 0.40 mg folic acid from enrollment to delivery.
  Arms: Folic acid

SUMMARY:
According to a national study in 2002, the prevalence of ID, IDA, and ID+IDA among pregnant women in China was 42.6%, 9.1%, and 61.7% respectively. A similar study in Hebei province at the same time showed that the prevalence of IDA among pregnant and lactating mothers was 46.39% and 47.21% respectively. There was a significant difference between urban and rural areas. Women living in rural areas had higher chances of having IDA (p<0.01). WHO and UNICEF recommend taking iron, folic acid and multiple micronutrients during pregnancy. However, we don't know much about their influence on maternal and infant health and their clinical effectiveness. Health Department of China recommends taking 400ug folic acid before pregnancy and during early pregnancy. But for various reasons, not all expecting mothers take this advice. Besides, we don't have a national level technical standard of how to take nutrition supplements during pregnancy. Therefore, it's crucial for us to study if iron/folic acid or folic acid only can prevent perinatal complications, as well as their influences on infant and toddler health.

The purpose of this study is to test whether taking iron/folic acid and folic acid only from early pregnancy until delivery will lower the chances of pregnancy complications, and to see how supplements affect gestation results. As well, it will evaluate a) whether taking iron supplement during pregnancy can prevent IDA during pregnancy; b) whether taking iron supplement can increase mother and fetus iron storage; and c) how mother's iron level affects newborn's iron level. We hope to understand nutrition conditions during pregnancy and investigate the relations between pregnancy diet and complications during pregnancy, weight gain during pregnancy, and newborn birth weight. We will evaluate the influence of taking iron and folic acid during pregnancy on the health of infants and toddlers.

DETAILED DESCRIPTION:
Iron deficiency (ID) is the world's most common single nutrient disorder, differentially affecting pregnant women and infants everywhere. The study was conducted in China, a rapidly developing country where ID often occurs among pregnant women and infants in the absence of generalized undernutrition. The study was a collaboration between Peking University First Hospital and three local hospitals (Sanhe Maternity and Child Health Care Center [MCHC], Sanhe General County Hospital, and Sanhe Hospital of Traditional Chinese Medicine). Eligible pregnant women were enrolled from June 2009 through December 2011 and randomized in a 1:1 ratio to receive iron and folic acid or folic acid only. The study protocol was approved by the institutional review board of Peking University First Hospital, Beijing, China. Women were recruited (n=2367) at their first prenatal visit at Sanhe MCHC. Those with uncomplicated singleton pregnancies and first prenatal visits ≤ 20 weeks gestation were invited to participate. Women were randomized and received 2 supplements: iron/placebo and folic acid. Project personnel instructed the participants to take two capsules per day (one of each kind of supplement) from enrollment to delivery. Participants received a 3-month supply of each supplement upon enrollment and at the second study visit (26-30 weeks). The number of doses received and consumed or missed was recorded by project personnel. The primary outcomes were maternal iron status at follow-up visits (26-30 weeks and 36-40 weeks), cord-blood iron status, and infant gestational age and birth weight. Data analysis compares pregnancy iron level between two study groups and how it relates to pregnancy outcomes, including pregnancy and delivery complications, preterm rate, perinatal death rate, and birth rate. Data analysis also includes evaluating pregnancy nutrition conditions and analyzing associations with weight changes during pregnancy, and rates of pregnancy diabetes, pregnancy high blood pressure, fetus growth restriction, low birth weight, and fetal macrosomia. Up to 75% of pregnant women worldwide are anemic, with about half due to ID. The public health implications of study findings could be profound.

ELIGIBILITY:
Inclusion Criteria:

* uncomplicated singleton pregnancy, first enrollment visit ≤ 20 weeks gestation -

Exclusion Criteria:

* < 18 years of age
* did not live in the county
* did not anticipate delivery at participating hospital
* were not mentally competent
* had a chronic health problem or hemoglobin < 100 g/L at the initial visit
* were taking iron at the time.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2367 (Actual)
Dates: Start 2009-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Maternal iron status at follow-up prenatal visit | 26-30 weeks
Maternal iron status at follow-up prenatal visit | 36-40 weeks

SECONDARY OUTCOMES:
Cord-blood iron status | delivery
Infant gestational age | delivery
Infant birth weight | delivery

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Gengli, MD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, China

REFERENCES:
- [Derived] Finkelstein JL, Cuthbert A, Weeks J, Venkatramanan S, Larvie DY, De-Regil LM, Garcia-Casal MN. Daily oral iron supplementation during pregnancy. Cochrane Database Syst Rev. 2024 Aug 15;8(8):CD004736. doi: 10.1002/14651858.CD004736.pub6. PMID 39145520
- [Derived] Zhao G, Xu G, Zhou M, Jiang Y, Richards B, Clark KM, Kaciroti N, Georgieff MK, Zhang Z, Tardif T, Li M, Lozoff B. Prenatal Iron Supplementation Reduces Maternal Anemia, Iron Deficiency, and Iron Deficiency Anemia in a Randomized Clinical Trial in Rural China, but Iron Deficiency Remains Widespread in Mothers and Neonates. J Nutr. 2015 Aug;145(8):1916-23. doi: 10.3945/jn.114.208678. Epub 2015 Jun 10. PMID 26063068